CLINICAL TRIAL: NCT00995423
Title: Comparison of the Efficacy and Safety of Paclitaxel-Eluting CoroflexTM Please Stent Versus Paclitaxel-Eluting Stent in Patients With Coronary Artery Disease
Brief Title: Comparison of Paclitaxel-Eluting Coroflex Please Stent Versus Paclitaxel-Eluting Stent
Acronym: PIPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Seung-Jung Park, CardioVascular Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-0497
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CoroflexTM (Active Comparator): highly flexible CoroflexTM Please-Stent features
  Interventions: Device: CoroflexTM Please
- TAXUS (Active Comparator): Paclitaxel-eluting stent
  Interventions: Device: Paclitaxel-eluting stent

INTERVENTIONS:
Device: CoroflexTM Please — highly flexible CoroflexTM Please-Stent
  Arms: CoroflexTM
Device: Paclitaxel-eluting stent — Paclitaxel-eluting stent
  Other Names: Taxus liberte
  Arms: TAXUS

SUMMARY:
The purpose of this study is to assess whether the outcome of treatment with CoroflexTM Please stent is not inferior to the outcome of treatment with TAXUS stent.

DETAILED DESCRIPTION:
To establish the effectiveness and the safety of coronary stenting with the newly developed paclitaxel-eluting balloon expandable stent (CoroflexTM Please stent, B. Bran, Melsungen, Germany), compared to the conventional paclitaxel-eluting balloon expandable stent (TAXUS stent, Boston scientific) in the treatment of coronary stenosis.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age
* Significant de novo coronary artery stenosis (>50% by visual estimation)
* Patients with stable (CCS class 1 to 4) or acute coronary syndromes (unstable angina pectoris Braunwald class IB, IC, IIB, IIC, IIIB, IIIC or NSTEMI) or patents with atypical chest pain or without symptoms but having documented myocardial ischemia, amenable to stent-assisted percutaneous coronary intervention
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications:

  * Heparin
  * Aspirin
  * Both Clopidogrel and TIclopidine
  * Sirolimus, paclitaxel
  * Stainless steel and/or
  * Contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled)
* Systemic (intravenous) Sirolimus or paclitaxel use within 12 months
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months
* Current known current platelet count <100,000 cells/mm3 or Hgb <10 g/dL
* An elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first 12 months post enrollment
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period
* Patients with EF<25%
* Cardiogenic shock at entry
* Acute MI patients within symptom onset < 12 hours needing primary angioplasty
* Creatinine level > 3.0mg/dL or dependence on dialysis
* Patients with left main stem stenosis (>50% by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
In-segment late lumen loss by quantitative coronary angiographic measurements | 9 months

SECONDARY OUTCOMES:
All Death | 12 months
Cardiac death | 12 months
Myocardial infarction | 12 month
Target vessel revascularization (all and ischemia-driven) | 12 month
Target lesion revascularization (all and ischemia-driven) | 12 months
Stent thrombosis (by ARC definition) | 12 months
In-stent late loss at 9 month angiographic follow-up | 12 months
Binary restenosis in both in-stent and in-segment | 9 month
Angiographic pattern of restenosis | 9 months
Procedural success defined as achievement of a final diameter stenosis of <30% by QCA using any percutaneous method, without the occurrence of death, Q wave MI, or repeat revascularization of the target lesion | during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (10):
- South Korea (10):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Chungnam National University Hospital, Daejeon
  - Asan Medical Center, Gangneung
  - Kwangju Christian Hospital, Kwangju
  - Hallym University Sacred Heart Hospital, Pyeongchon
  - Asan Medical Center, Seoul
  - Hangang Sacred Heart Hospital, Seoul
  - Seoul Veterans Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan